CLINICAL TRIAL: NCT00228917
Title: Assess Reactogenicity & Safety of a Booster of Either Tritanrix-HepB/Hib-MenAC or Tritanrix-HepB/Hiberix Given (Single-blind) at 15-18 (Philippines)/15-24 Mths (Thailand) & a Dose of Mencevax ACWY at 24-30 Mths (Open Label)
Brief Title: Safety Study of Tritanrix-HepB/Hib-MenAC, Tritanrix-HepB/Hiberix, and Mencevax ACWY Vaccines in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103812; 104171 (Other: GSK)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Whole Cell Pertussis; Tetanus; Hepatitis B; Diphtheria; Haemophilus Influenzae Type b; Diphtheria-Tetanus-Pertussis-Hepatitis B-Haemophilus Influenzae Type b-Neisseria Meningitidis Vaccin
Keywords: Hib & Neisseria meningitidis serogroups A & C diseases
MeSH Terms: conditions — Tetanus; Hepatitis B; Diphtheria; Haemophilus Infections | interventions — PsACWY vaccine

STUDY DESIGN:
Who Masked: Participant

ARMS (8):
- ACAC_Thailand Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine in the primary study ( NCT00317187) are boosted in the current study with one dose of the same vaccines at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age
  Interventions: Biological: Tritanrix-HepB/Hib-MenAC
- ACHibPS_Thailand Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine in the primary study (NCT00317187) are boosted in the current study with one dose of Tritanrix-HepB/Hiberix at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Tritanrix-HepB/Hiberix; Biological: Mencevax-ACWY
- HibACPS_Thailand Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317187) are boosted in the current study with one dose of Trianrix-Hepb co-administrated with Hib-MenAC-TT vaccine at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Tritanrix-HepB/Hib-MenAC; Biological: Mencevax-ACWY
- HibHibPS_Thailand Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317187) are boosted in the current study with one dose of the same vaccine at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Tritanrix-HepB/Hiberix; Biological: Mencevax-ACWY
- ACAC_Philippines Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine in the primary study (NCT00317135) are boosted in the current study with one dose of the same vaccines at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age
  Interventions: Biological: Tritanrix-HepB/Hib-MenAC
- ACHibPS_Philippines Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine in the primary study (NCT00317135) are boosted in the current study with one dose of Tritanrix-HepB/Hiberix at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Tritanrix-HepB/Hiberix; Biological: Mencevax-ACWY
- HibACPS_Philippines Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317135) are boosted in the current study with one dose of Trianrix-Hepb co-administrated with Hib-MenAC-TT vaccine at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Tritanrix-HepB/Hib-MenAC; Biological: Mencevax-ACWY
- HibHibPS_Philippines Group (Experimental): Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317135) are boosted in the current study with one dose of the same vaccine at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Tritanrix-HepB/Hiberix; Biological: Mencevax-ACWY

INTERVENTIONS:
Biological: Tritanrix-HepB/Hib-MenAC — Combined Diphtheria, Tetanus, Whole Cell Pertussis, Hepatitis B, Haemophilus influenzae Type b meningococcal AC-tetanus toxoid conjugate Vaccine
  Arms: ACAC_Philippines Group; ACAC_Thailand Group; HibACPS_Philippines Group; HibACPS_Thailand Group
Biological: Tritanrix-HepB/Hiberix — Combined Diphtheria, Tetanus, Whole Cell Pertussis, Hepatitis B Vaccine, Haemophilus influenzae type b conjugate vaccine
  Arms: ACHibPS_Philippines Group; ACHibPS_Thailand Group; HibHibPS_Philippines Group; HibHibPS_Thailand Group
Biological: Mencevax-ACWY — Meningococcal Serogroups A, C, W-135 and Y Vaccine
  Arms: ACHibPS_Philippines Group; ACHibPS_Thailand Group; HibACPS_Philippines Group; HibACPS_Thailand Group; HibHibPS_Philippines Group; HibHibPS_Thailand Group

SUMMARY:
This study will be conducted in two stages. In the diphtheria, tetanus, pertussis (DTP) booster phase, subjects will receive a booster dose of Tritanrix-HepB/Hib-MenAC or Tritanrix-HepB/Hiberix (active control) at 15 to 18 or 24 months in a single-blind manner so that the subjects' parents will not know which vaccine was administered to their child. In the Mencevax ACWY phase at 24-30 months, a dose of Mencevax ACWY will be given in an open manner to only those subjects who received less than 4 doses of Tritanrix-HepB/Hib-MenAC. No blood samples will be taken in this safety study.

DETAILED DESCRIPTION:
Subjects previously primed with Tritanrix-HepB/Hib-MenAC will receive Tritanrix-HepB/Hib-MenAC or Tritanrix-HepB/Hiberix vaccine (at 15-18/24 m), respectively, without or with Mencevax ACWY vaccine at 24 to 30 months of age. Subjects previously primed with Tritanrix-HepB/Hiberix will receive Tritanrix-HepB/Hib-MenAC or Tritanrix-HepB/Hiberix vaccine (at 15-18/24 m) with Mencevax ACWY vaccine at 24 to 30 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the parent or guardian of a healthy male or female child between, and including 15 and 18 months age (Philippines)/ 15 and 24 months age (Thailand) at the time of vaccination and who have previously received a 3-dose primary vaccination in the studies DTPwHB/HibMenAC-TT-004 (CPMS No. 759346/004) or DTPW-HBV=HIB-MENAC-TT-013 (eTrack No. 100791).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the vaccination, or planned use during the study period.
* Chronic administration (> than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of vaccination. Note: Oral poliovirus vaccine can be given concomitantly.
* Booster vaccination against diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b (Hib) and/or meningococcal serogroups A and C disease, after the date of the study conclusion visit of the primary vaccination study.

Ages: 427 Days to 577 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 798 (Actual)
Dates: Start 2005-06-16 (Actual); Primary Completion 2006-01-20 (Actual); Study Completion 2006-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, City of Muntinlupa, Philippines
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 103812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 103812 are summarised with study 104727 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 103812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103812 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- ACAC_Thailand Group: Subjects vaccinated with 3 doses of Tritanrix-HepB co-administrated with Hib-MenAC-TT vaccine in the primary study (NCT00317187) were boosted in the current study with one dose of the same vaccines at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age
- ACHibPS_Thailand Group: Subjects vaccinated with 3 doses of Trianrix-HepB coadministrated with Hib-MenAC-TT vaccine in the primary study (NCT00317187) were boosted in the current study with one dose of Tritanrix HepB/Hiberix at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
- HibACPS_Thailand Group: Subjects vaccinated with 3 doses of Tritanrix HepB/Hiberix vaccine in the primary study (NCT00317187) were boosted in the current study with one dose of Trianrix-HepB coadministrated with Hib-MenAC-TT vaccine at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
- HibHibPS_Thailand Group: Subjects vaccinated with 3 doses of Tritanrix HepB/Hiberix vaccine in the primary study (NCT00317187) were boosted in the current study with one dose of the same vaccine at 15 to 24 months (Thailand) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
- ACAC_Philippines Group: Subjects vaccinated with 3 doses of Tritanrix HepB coadministrated with Hib-MenAC-TT vaccine in the primary study (NCT00317135) were boosted in the current study with one dose of the same vaccines at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age
- ACHibPS_Philippines Group: Subjects vaccinated with 3 doses of Trianrix-Hepb co-administrated with Mencevax vaccine in the primary study (NCT00317135) were boosted in the current study with one dose of Tritanrix-HepB/Hiberix at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
- HibACPS_Philippines Group: Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317135) were boosted in the current study with one dose of Trianrix-Hepb co-administrated with Hib-MenAC-TT vaccine at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
- HibHibPS_Philippines Group: Subjects vaccinated with 3 doses of Tritanrix HepB/Hiberix vaccine in the primary study (NCT00317135) were boosted in the current study with one dose of the same vaccine at 15 to 18 months (Philippines) of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
Period: Overall Study
Arm/Group | ACAC_Thailand Group | ACHibPS_Thailand Group | HibACPS_Thailand Group | HibHibPS_Thailand Group | ACAC_Philippines Group | ACHibPS_Philippines Group | HibACPS_Philippines Group | HibHibPS_Philippines Group
Started | 193 | 96 | 65 | 33 | 205 | 104 | 69 | 33
Completed | 193 | 96 | 65 | 33 | 205 | 102 | 69 | 33
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Total: Total of all reporting groups
Arm/Group | ACAC_Thailand Group | ACHibPS_Thailand Group | HibACPS_Thailand Group | HibHibPS_Thailand Group | ACAC_Philippines Group | ACHibPS_Philippines Group | HibACPS_Philippines Group | HibHibPS_Philippines Group | Total
Number analyzed (Participants) | 193 | 96 | 65 | 33 | 205 | 104 | 69 | 33 | 798
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.7 (0.7) | 17.8 (0.71) | 17.7 (0.78) | 17.6 (0.7) | 17.1 (0.78) | 17.2 (0.79) | 17.2 (0.93) | 17 (0.77) | 17.59 (0.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 45 | 32 | 18 | 107 | 56 | 29 | 16 | 399
  Male | 97 | 51 | 33 | 15 | 98 | 48 | 40 | 17 | 399

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Fever >39°C (Rectal Route).
Description: Among solicited general symptoms fever [defined as rectal temperature equal to or above (≥) 38 degrees Celsius (°C )] was assessed, post vaccination. Grade 3 fever = fever > 39.0 °C.
Time Frame: During the 4-day (Day 0-3) follow-up period after booster vaccination
Population: This analysis was performed on Booster Total Vaccinated cohort which included all subjects who have received three doses according to protocol in the primary vaccination course (primary vaccination studies) and who have received the booster vaccine dose according to protocol,only taking into account those subjects who returned their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | ACAC_Thailand Group | ACHibPS_Thailand Group | HibACPS_Thailand Group | HibHibPS_Thailand Group | ACAC_Philippines Group | ACHibPS_Philippines Group | HibACPS_Philippines Group | HibHibPS_Philippines Group
Number analyzed (Participants) | 193 | 96 | 65 | 33 | 205 | 102 | 69 | 33
Participants | 22 | 8 | 5 | 3 | 40 | 24 | 17 | 6

2. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms, Other Than Fever > 39.0°C
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period after vaccination
Population: This analysis was performed on the Booster Total Vaccinated cohort included all subjects who have received three doses according to protocol in the primary vaccination course (primary vaccination studies) and who have received the booster vaccine dose according to protocol,only taking into account those subjects who returned their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | ACAC_Thailand Group | ACHibPS_Thailand Group | HibACPS_Thailand Group | HibHibPS_Thailand Group | ACAC_Philippines Group | ACHibPS_Philippines Group | HibACPS_Philippines Group | HibHibPS_Philippines Group
Number analyzed (Participants) | 193 | 96 | 65 | 33 | 205 | 102 | 69 | 33
Participants
  Any Drowsiness | 113 | 63 | 41 | 17 | 53 | 33 | 23 | 8
  Grade 3 Drowsiness | 6 | 0 | 0 | 0 | 3 | 0 | 2 | 1
  Related Drowsiness | 110 | 63 | 41 | 17 | 16 | 7 | 4 | 1
  Any Irritability | 149 | 75 | 53 | 26 | 116 | 59 | 39 | 17
  Grade 3 Irritability | 21 | 3 | 7 | 5 | 4 | 2 | 1 | 1
  Related Irritability | 146 | 74 | 53 | 26 | 29 | 15 | 6 | 4
  Any Loss of appetite | 98 | 46 | 33 | 15 | 72 | 40 | 24 | 6
  Grade 3 Loss of appetite | 7 | 1 | 2 | 1 | 1 | 0 | 0 | 0
  Related Loss of appetite | 96 | 46 | 33 | 15 | 18 | 10 | 2 | 1
  Fever ≥ 38.5°C | 55 | 24 | 19 | 7 | 80 | 41 | 35 | 10
  Fever ≥ 40.0°C | 1 | 0 | 2 | 1 | 5 | 2 | 3 | 1
  Related Fever | 112 | 57 | 47 | 18 | 34 | 21 | 5 | 4

3. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-3) follow-up period after booster vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | ACAC_Thailand Group | ACHibPS_Thailand Group | HibACPS_Thailand Group | HibHibPS_Thailand Group | ACAC_Philippines Group | ACHibPS_Philippines Group | HibACPS_Philippines Group | HibHibPS_Philippines Group
Number analyzed (Participants) | 193 | 96 | 65 | 33 | 205 | 102 | 69 | 33
Subjects
  Any Pain | 168 | 78 | 55 | 26 | 151 | 69 | 49 | 22
  Grade 3 Pain | 57 | 14 | 12 | 4 | 42 | 13 | 22 | 8
  Any Redness | 99 | 33 | 33 | 16 | 40 | 33 | 21 | 9
  Grade 3 Redness | 12 | 0 | 3 | 1 | 1 | 0 | 1 | 0
  Any Swelling | 95 | 33 | 33 | 14 | 51 | 32 | 21 | 10
  Grade 3 Swelling | 18 | 5 | 8 | 1 | 10 | 6 | 3 | 0

4. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-30) following booster vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | ACAC_Thailand Group | ACHibPS_Thailand Group | HibACPS_Thailand Group | HibHibPS_Thailand Group | ACAC_Philippines Group | ACHibPS_Philippines Group | HibACPS_Philippines Group | HibHibPS_Philippines Group
Number analyzed (Participants) | 193 | 96 | 65 | 33 | 205 | 102 | 69 | 33
Subjects | 64 | 23 | 24 | 9 | 53 | 33 | 16 | 6

5. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From 15 to 18 months or 15 to 24 months of age and up to 25 to 31 months of age post vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | ACAC_Thailand Group | ACHibPS_Thailand Group | HibACPS_Thailand Group | HibHibPS_Thailand Group | ACAC_Philippines Group | ACHibPS_Philippines Group | HibACPS_Philippines Group | HibHibPS_Philippines Group
Number analyzed (Participants) | 193 | 96 | 65 | 33 | 205 | 102 | 69 | 33
Subjects | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms during the 4-day(Day 0-3)follow-up period after vaccination. Unsolicited AEs during the 31-day(Day 0-30)follow-up period after vaccination.SAEs from 15 to 18 months/15 to 24 months of age and up to 25 to 31 months of age(i.e a duration of Minimum of 6 months and a maximum of 16 months per subject(depending on the study group,on the recommended national vaccination schedule and on how the study will be organized at the different centers by the investigators)
Description: Detailed analysis (i.e solicited and unsolicited merge analysis for other adverse event section as well as medical coding for this adverse event section) was only performed on the pooled groups
Groups:
- ACAC Group: Subjects from both ACAC_Thailand and ACAC_Philippines groups
- ACHibPS Group: Subjects from both ACHibPS_Thailand and ACHibPS_Philippines groups
- HibACPS Group: Subjects from both HibACPS_Thailand and HibACPS_Philippines groups
- HibHibPS Group: Subjects from both HibHibPS _Thailand and HibHibPS _Philippines groups
Arm/Group | ACAC Group | ACHibPS Group | HibACPS Group | HibHibPS Group
All-Cause Mortality (participants affected / at risk) | 0/398 | 0/200 | 0/134 | 0/66
Serious Adverse Events (participants affected / at risk) | 5/398 | 1/200 | 0/134 | 0/66
Other Adverse Events (participants affected / at risk) | 376/398 | 181/200 | 129/134 | 60/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACAC Group (N=398) | ACHibPS Group (N=200) | HibACPS Group (N=134) | HibHibPS Group (N=66)
Febrile convulsion (Nervous system disorders) | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Measles (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACAC Group (N=398) | ACHibPS Group (N=200) | HibACPS Group (N=134) | HibHibPS Group (N=66)
Pain (General disorders) | 319 | 147 | 104 | 48
Swelling (General disorders) | 146 | 65 | 54 | 24
Pyrexia (General disorders) | 272 | 126 | 99 | 41
Upper respiratory tract infection (Infections and infestations) | 36 | 16 | 9 | 4
Irritability (Psychiatric disorders) | 265 | 134 | 92 | 43
Decreased appetite (Metabolism and nutrition disorders) | 170 | 86 | 57 | 21
Erythema (Skin and subcutaneous tissue disorders) | 139 | 66 | 54 | 25
Nasopharyngitis (Infections and infestations) | 10 | 4 | 8 | 2
Somnolence (Nervous system disorders) | 166 | 96 | 64 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.